CLINICAL TRIAL: NCT04223102
Title: Rectal Microbiome Variability Among Rectal Cancer Cohorts Including Complete Clinical Responders, Pathologic Responders, and Early Recurrence
Brief Title: Microbiome and Rectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00040924
Record Dates: First submitted 2019-11-12; First posted 2020-01-10 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Rectal Cancer; Locally Advanced Malignant Neoplasm
MeSH Terms: conditions — Rectal Neoplasms | interventions — Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tissue collection (Other): Tissue collection
  Interventions: Procedure: Tissue collection

INTERVENTIONS:
Procedure: Tissue collection — A flexible sigmoidoscopy is a procedure in which a flexible tubularized camera approximately 1 cm in diameter is inserted into the anus and advanced proximally to the sigmoid colon (approximately 20 cm). At that time a rectal biopsy of the tumor will be obtained as well as a sample from >5cm proximal to the tumor, with a separate biopsy forcep. Tattoo injection, as standard of care, will be performed within 1 cm distal to the tumor to identify the location in the future or for surgical intervention. If there is inability to get proximal to the tumor then a location at least 5 cm adjacent in any direction will be sufficient so long as it is grossly normal appearing.

SUMMARY:
The purpose of our study is to determine if an association exists between the microbiome of those with rectal adenocarcinoma who are complete pathologic responders and those who have a partial or no response to neoadjuvant therapy.

DETAILED DESCRIPTION:
This study will help to further elucidate the association of bacteria with rectal cancer, while also characterizing the genes associated with that risk. Furthermore it will attempt to better understand which patients may have an optimal response to neoadjuvant chemoradiation allowing for possible predictive metagenomics evaluation, investigators may be able to augment treatments as well as provide recommendations for the success and cost effectiveness of cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Locally Advanced Rectal Adenocarcinoma (T3)
* Standard 5FU based chemoradiation
* Total Neoadjuvant Therapy per OPRA protocol guidelines

Exclusion Criteria:

* Age < 18 years
* Stage I or Stage IV rectal adenocarcinoma
* Rectal cancer other than adenocarcinoma
* Genetically associated cancer (HNPCC, FAP etc.) or highly suspicious for genetically associated cancer
* Prior history of rectal adenocarcinoma (i.e. recurrent colorectal adenocarcinoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
16s rRNA gene sequencing to study bacterial phylogeny and taxonomy | 5 years
  16s rRNA sequencing from biopsy specimens

SECONDARY OUTCOMES:
rectal microbiota to study bacteria strains | 5 years
  rectal microbiota - bacteria strains from biopsy specimens

CONTACTS AND LOCATIONS:
Overall Officials: James R Williams, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida
  - University of South Florida, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NIH HMP Working Group; Peterson J, Garges S, Giovanni M, McInnes P, Wang L, Schloss JA, Bonazzi V, McEwen JE, Wetterstrand KA, Deal C, Baker CC, Di Francesco V, Howcroft TK, Karp RW, Lunsford RD, Wellington CR, Belachew T, Wright M, Giblin C, David H, Mills M, Salomon R, Mullins C, Akolkar B, Begg L, Davis C, Grandison L, Humble M, Khalsa J, Little AR, Peavy H, Pontzer C, Portnoy M, Sayre MH, Starke-Reed P, Zakhari S, Read J, Watson B, Guyer M. The NIH Human Microbiome Project. Genome Res. 2009 Dec;19(12):2317-23. doi: 10.1101/gr.096651.109. Epub 2009 Oct 9. PMID 19819907
- [Background] Smith JJ, Chow OS, Gollub MJ, Nash GM, Temple LK, Weiser MR, Guillem JG, Paty PB, Avila K, Garcia-Aguilar J; Rectal Cancer Consortium. Organ Preservation in Rectal Adenocarcinoma: a phase II randomized controlled trial evaluating 3-year disease-free survival in patients with locally advanced rectal cancer treated with chemoradiation plus induction or consolidation chemotherapy, and total mesorectal excision or nonoperative management. BMC Cancer. 2015 Oct 23;15:767. doi: 10.1186/s12885-015-1632-z. PMID 26497495
- [Background] Maas M, Nelemans PJ, Valentini V, Das P, Rodel C, Kuo LJ, Calvo FA, Garcia-Aguilar J, Glynne-Jones R, Haustermans K, Mohiuddin M, Pucciarelli S, Small W Jr, Suarez J, Theodoropoulos G, Biondo S, Beets-Tan RG, Beets GL. Long-term outcome in patients with a pathological complete response after chemoradiation for rectal cancer: a pooled analysis of individual patient data. Lancet Oncol. 2010 Sep;11(9):835-44. doi: 10.1016/S1470-2045(10)70172-8. Epub 2010 Aug 6. PMID 20692872
- [Background] Smith JD, Ruby JA, Goodman KA, Saltz LB, Guillem JG, Weiser MR, Temple LK, Nash GM, Paty PB. Nonoperative management of rectal cancer with complete clinical response after neoadjuvant therapy. Ann Surg. 2012 Dec;256(6):965-72. doi: 10.1097/SLA.0b013e3182759f1c. PMID 23154394
- [Background] Gerassy-Vainberg S, Blatt A, Danin-Poleg Y, Gershovich K, Sabo E, Nevelsky A, Daniel S, Dahan A, Ziv O, Dheer R, Abreu MT, Koren O, Kashi Y, Chowers Y. Radiation induces proinflammatory dysbiosis: transmission of inflammatory susceptibility by host cytokine induction. Gut. 2018 Jan;67(1):97-107. doi: 10.1136/gutjnl-2017-313789. Epub 2017 Apr 24. PMID 28438965
- [Background] Araujo-Perez F, McCoy AN, Okechukwu C, Carroll IM, Smith KM, Jeremiah K, Sandler RS, Asher GN, Keku TO. Differences in microbial signatures between rectal mucosal biopsies and rectal swabs. Gut Microbes. 2012 Nov-Dec;3(6):530-5. doi: 10.4161/gmic.22157. Epub 2012 Oct 11. PMID 23060016
- [Result] Peters BA, Wu J, Pei Z, Yang L, Purdue MP, Freedman ND, Jacobs EJ, Gapstur SM, Hayes RB, Ahn J. Oral Microbiome Composition Reflects Prospective Risk for Esophageal Cancers. Cancer Res. 2017 Dec 1;77(23):6777-6787. doi: 10.1158/0008-5472.CAN-17-1296. PMID 29196415
- [Result] Sanapareddy N, Legge RM, Jovov B, McCoy A, Burcal L, Araujo-Perez F, Randall TA, Galanko J, Benson A, Sandler RS, Rawls JF, Abdo Z, Fodor AA, Keku TO. Increased rectal microbial richness is associated with the presence of colorectal adenomas in humans. ISME J. 2012 Oct;6(10):1858-68. doi: 10.1038/ismej.2012.43. Epub 2012 May 24. PMID 22622349
- [Result] Xu K, Jiang B. Analysis of Mucosa-Associated Microbiota in Colorectal Cancer. Med Sci Monit. 2017 Sep 14;23:4422-4430. doi: 10.12659/msm.904220. PMID 28904330
- [Result] Kwong TNY, Wang X, Nakatsu G, Chow TC, Tipoe T, Dai RZW, Tsoi KKK, Wong MCS, Tse G, Chan MTV, Chan FKL, Ng SC, Wu JCY, Wu WKK, Yu J, Sung JJY, Wong SH. Association Between Bacteremia From Specific Microbes and Subsequent Diagnosis of Colorectal Cancer. Gastroenterology. 2018 Aug;155(2):383-390.e8. doi: 10.1053/j.gastro.2018.04.028. Epub 2018 May 3. PMID 29729257
- [Result] Kasai C, Sugimoto K, Moritani I, Tanaka J, Oya Y, Inoue H, Tameda M, Shiraki K, Ito M, Takei Y, Takase K. Comparison of human gut microbiota in control subjects and patients with colorectal carcinoma in adenoma: Terminal restriction fragment length polymorphism and next-generation sequencing analyses. Oncol Rep. 2016 Jan;35(1):325-33. doi: 10.3892/or.2015.4398. Epub 2015 Nov 4. PMID 26549775
- [Result] Yoon H, Kim N, Park JH, Kim YS, Lee J, Kim HW, Choi YJ, Shin CM, Park YS, Lee DH, Jung HC. Comparisons of Gut Microbiota Among Healthy Control, Patients With Conventional Adenoma, Sessile Serrated Adenoma, and Colorectal Cancer. J Cancer Prev. 2017 Jun;22(2):108-114. doi: 10.15430/JCP.2017.22.2.108. Epub 2017 Jun 30. PMID 28698865
- [Result] Ahn J, Sinha R, Pei Z, Dominianni C, Wu J, Shi J, Goedert JJ, Hayes RB, Yang L. Human gut microbiome and risk for colorectal cancer. J Natl Cancer Inst. 2013 Dec 18;105(24):1907-11. doi: 10.1093/jnci/djt300. Epub 2013 Dec 6. PMID 24316595
- [Result] Chen W, Liu F, Ling Z, Tong X, Xiang C. Human intestinal lumen and mucosa-associated microbiota in patients with colorectal cancer. PLoS One. 2012;7(6):e39743. doi: 10.1371/journal.pone.0039743. Epub 2012 Jun 28. PMID 22761885
- [Result] Jones RB, Zhu X, Moan E, Murff HJ, Ness RM, Seidner DL, Sun S, Yu C, Dai Q, Fodor AA, Azcarate-Peril MA, Shrubsole MJ. Inter-niche and inter-individual variation in gut microbial community assessment using stool, rectal swab, and mucosal samples. Sci Rep. 2018 Mar 7;8(1):4139. doi: 10.1038/s41598-018-22408-4. PMID 29515151
- [Result] Mandal P. Molecular mechanistic pathway of colorectal carcinogenesis associated with intestinal microbiota. Anaerobe. 2018 Feb;49:63-70. doi: 10.1016/j.anaerobe.2017.12.008. Epub 2017 Dec 19. PMID 29277623
- [Result] Chen GY. The Role of the Gut Microbiome in Colorectal Cancer. Clin Colon Rectal Surg. 2018 May;31(3):192-198. doi: 10.1055/s-0037-1602239. Epub 2018 Apr 1. PMID 29720905
- [Result] Flemer B, Lynch DB, Brown JM, Jeffery IB, Ryan FJ, Claesson MJ, O'Riordain M, Shanahan F, O'Toole PW. Tumour-associated and non-tumour-associated microbiota in colorectal cancer. Gut. 2017 Apr;66(4):633-643. doi: 10.1136/gutjnl-2015-309595. Epub 2016 Mar 18. PMID 26992426
- [Result] Mima K, Sukawa Y, Nishihara R, Qian ZR, Yamauchi M, Inamura K, Kim SA, Masuda A, Nowak JA, Nosho K, Kostic AD, Giannakis M, Watanabe H, Bullman S, Milner DA, Harris CC, Giovannucci E, Garraway LA, Freeman GJ, Dranoff G, Chan AT, Garrett WS, Huttenhower C, Fuchs CS, Ogino S. Fusobacterium nucleatum and T Cells in Colorectal Carcinoma. JAMA Oncol. 2015 Aug;1(5):653-61. doi: 10.1001/jamaoncol.2015.1377. PMID 26181352
- [Result] Mima K, Nishihara R, Qian ZR, Cao Y, Sukawa Y, Nowak JA, Yang J, Dou R, Masugi Y, Song M, Kostic AD, Giannakis M, Bullman S, Milner DA, Baba H, Giovannucci EL, Garraway LA, Freeman GJ, Dranoff G, Garrett WS, Huttenhower C, Meyerson M, Meyerhardt JA, Chan AT, Fuchs CS, Ogino S. Fusobacterium nucleatum in colorectal carcinoma tissue and patient prognosis. Gut. 2016 Dec;65(12):1973-1980. doi: 10.1136/gutjnl-2015-310101. Epub 2015 Aug 26. PMID 26311717
- [Result] Liu L, Tabung FK, Zhang X, Nowak JA, Qian ZR, Hamada T, Nevo D, Bullman S, Mima K, Kosumi K, da Silva A, Song M, Cao Y, Twombly TS, Shi Y, Liu H, Gu M, Koh H, Li W, Du C, Chen Y, Li C, Li W, Mehta RS, Wu K, Wang M, Kostic AD, Giannakis M, Garrett WS, Hutthenhower C, Chan AT, Fuchs CS, Nishihara R, Ogino S, Giovannucci EL. Diets That Promote Colon Inflammation Associate With Risk of Colorectal Carcinomas That Contain Fusobacterium nucleatum. Clin Gastroenterol Hepatol. 2018 Oct;16(10):1622-1631.e3. doi: 10.1016/j.cgh.2018.04.030. Epub 2018 Apr 24. PMID 29702299
- [Result] McCoy AN, Araujo-Perez F, Azcarate-Peril A, Yeh JJ, Sandler RS, Keku TO. Fusobacterium is associated with colorectal adenomas. PLoS One. 2013;8(1):e53653. doi: 10.1371/journal.pone.0053653. Epub 2013 Jan 15. PMID 23335968
- [Result] Flanagan L, Schmid J, Ebert M, Soucek P, Kunicka T, Liska V, Bruha J, Neary P, Dezeeuw N, Tommasino M, Jenab M, Prehn JH, Hughes DJ. Fusobacterium nucleatum associates with stages of colorectal neoplasia development, colorectal cancer and disease outcome. Eur J Clin Microbiol Infect Dis. 2014 Aug;33(8):1381-90. doi: 10.1007/s10096-014-2081-3. Epub 2014 Mar 6. PMID 24599709
- [Result] Mima K, Cao Y, Chan AT, Qian ZR, Nowak JA, Masugi Y, Shi Y, Song M, da Silva A, Gu M, Li W, Hamada T, Kosumi K, Hanyuda A, Liu L, Kostic AD, Giannakis M, Bullman S, Brennan CA, Milner DA, Baba H, Garraway LA, Meyerhardt JA, Garrett WS, Huttenhower C, Meyerson M, Giovannucci EL, Fuchs CS, Nishihara R, Ogino S. Fusobacterium nucleatum in Colorectal Carcinoma Tissue According to Tumor Location. Clin Transl Gastroenterol. 2016 Nov 3;7(11):e200. doi: 10.1038/ctg.2016.53. PMID 27811909
- [Result] Yang Y, Weng W, Peng J, Hong L, Yang L, Toiyama Y, Gao R, Liu M, Yin M, Pan C, Li H, Guo B, Zhu Q, Wei Q, Moyer MP, Wang P, Cai S, Goel A, Qin H, Ma Y. Fusobacterium nucleatum Increases Proliferation of Colorectal Cancer Cells and Tumor Development in Mice by Activating Toll-Like Receptor 4 Signaling to Nuclear Factor-kappaB, and Up-regulating Expression of MicroRNA-21. Gastroenterology. 2017 Mar;152(4):851-866.e24. doi: 10.1053/j.gastro.2016.11.018. Epub 2016 Nov 19. PMID 27876571
- [Result] Kostic AD, Chun E, Robertson L, Glickman JN, Gallini CA, Michaud M, Clancy TE, Chung DC, Lochhead P, Hold GL, El-Omar EM, Brenner D, Fuchs CS, Meyerson M, Garrett WS. Fusobacterium nucleatum potentiates intestinal tumorigenesis and modulates the tumor-immune microenvironment. Cell Host Microbe. 2013 Aug 14;14(2):207-15. doi: 10.1016/j.chom.2013.07.007. PMID 23954159
- [Result] Wong SH, Kwong TNY, Chow TC, Luk AKC, Dai RZW, Nakatsu G, Lam TYT, Zhang L, Wu JCY, Chan FKL, Ng SSM, Wong MCS, Ng SC, Wu WKK, Yu J, Sung JJY. Quantitation of faecal Fusobacterium improves faecal immunochemical test in detecting advanced colorectal neoplasia. Gut. 2017 Aug;66(8):1441-1448. doi: 10.1136/gutjnl-2016-312766. Epub 2016 Oct 24. PMID 27797940
- [Result] Sears CL. The who, where and how of fusobacteria and colon cancer. Elife. 2018 Mar 13;7:e28434. doi: 10.7554/eLife.28434. PMID 29533185
- [Result] Abed J, Maalouf N, Parhi L, Chaushu S, Mandelboim O, Bachrach G. Tumor Targeting by Fusobacterium nucleatum: A Pilot Study and Future Perspectives. Front Cell Infect Microbiol. 2017 Jun 30;7:295. doi: 10.3389/fcimb.2017.00295. eCollection 2017. PMID 28713780
- [Result] Rubinstein MR, Wang X, Liu W, Hao Y, Cai G, Han YW. Fusobacterium nucleatum promotes colorectal carcinogenesis by modulating E-cadherin/beta-catenin signaling via its FadA adhesin. Cell Host Microbe. 2013 Aug 14;14(2):195-206. doi: 10.1016/j.chom.2013.07.012. PMID 23954158
- [Result] Chen Y, Peng Y, Yu J, Chen T, Wu Y, Shi L, Li Q, Wu J, Fu X. Invasive Fusobacterium nucleatum activates beta-catenin signaling in colorectal cancer via a TLR4/P-PAK1 cascade. Oncotarget. 2017 May 9;8(19):31802-31814. doi: 10.18632/oncotarget.15992. PMID 28423670
- [Result] Bullman S, Pedamallu CS, Sicinska E, Clancy TE, Zhang X, Cai D, Neuberg D, Huang K, Guevara F, Nelson T, Chipashvili O, Hagan T, Walker M, Ramachandran A, Diosdado B, Serna G, Mulet N, Landolfi S, Ramon Y Cajal S, Fasani R, Aguirre AJ, Ng K, Elez E, Ogino S, Tabernero J, Fuchs CS, Hahn WC, Nuciforo P, Meyerson M. Analysis of Fusobacterium persistence and antibiotic response in colorectal cancer. Science. 2017 Dec 15;358(6369):1443-1448. doi: 10.1126/science.aal5240. Epub 2017 Nov 23. PMID 29170280
- [Result] Wirbel J, Pyl PT, Kartal E, Zych K, Kashani A, Milanese A, Fleck JS, Voigt AY, Palleja A, Ponnudurai R, Sunagawa S, Coelho LP, Schrotz-King P, Vogtmann E, Habermann N, Nimeus E, Thomas AM, Manghi P, Gandini S, Serrano D, Mizutani S, Shiroma H, Shiba S, Shibata T, Yachida S, Yamada T, Waldron L, Naccarati A, Segata N, Sinha R, Ulrich CM, Brenner H, Arumugam M, Bork P, Zeller G. Meta-analysis of fecal metagenomes reveals global microbial signatures that are specific for colorectal cancer. Nat Med. 2019 Apr;25(4):679-689. doi: 10.1038/s41591-019-0406-6. Epub 2019 Apr 1. PMID 30936547
- [Result] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751
- [Result] Thomas AM, Jesus EC, Lopes A, Aguiar S Jr, Begnami MD, Rocha RM, Carpinetti PA, Camargo AA, Hoffmann C, Freitas HC, Silva IT, Nunes DN, Setubal JC, Dias-Neto E. Tissue-Associated Bacterial Alterations in Rectal Carcinoma Patients Revealed by 16S rRNA Community Profiling. Front Cell Infect Microbiol. 2016 Dec 9;6:179. doi: 10.3389/fcimb.2016.00179. eCollection 2016. PMID 28018861